CLINICAL TRIAL: NCT00003751
Title: Phase II Study of Penicillamine and Reduction of Copper for Angiosuppressive Therapy of Adults With Newly Diagnosed Glioblastoma
Brief Title: Penicillamine, Low Copper Diet, and Radiation Therapy in Treating Patients With Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NABTT-9704 CDR0000066872; U01CA062475 (NIH); NABTT-9704; JHOC-NABTT-9704
Record Dates: First submitted 1999-11-01; First posted 2004-08-18 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Penicillamine; Radiotherapy

INTERVENTIONS:
Drug: penicillamine
Radiation: radiation therapy

SUMMARY:
RATIONALE: Penicillamine may stop the growth of glioblastomas by stopping blood flow to the tumor. A diet low in copper may interfere with the growth of brain tumor cells. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining these therapies may be effective in treating glioblastoma.

PURPOSE: Phase II trial to study the effectiveness of penicillamine, a low copper diet, and radiation therapy in treating patients who have newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of penicillamine and copper reduction on survival and time to progression in adults with newly diagnosed glioblastoma. II. Determine the effect of penicillamine on the reduction of serum copper in these patients. III. Determine whether penicillamine reduces the tumor volume, vascularity, invasion, and edema in these patients.

OUTLINE: Patients receive oral penicillamine on the following schedule: Week 1: once daily Week 2: two times daily Week 3: three times daily Week 4: four times daily Week 5 to end of study: increased dose four times daily. Patients also receive oral pyridoxine daily and maintain a low copper diet (no greater than 0.5 mg/day). This regimen is continued for up to 2 years in the absence of disease progression or unacceptable toxicity. Radiotherapy is administered over 6 weeks, beginning on day 1 of penicillamine therapy. Patients are followed every month (with MRI every 2 months) until death.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven supratentorial grade IV astrocytoma (glioblastoma multiforme)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: At least 2 months Hematopoietic: WBC at least 3000/mm3 Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10.0 g/dL No serious blood dyscrasias Hepatic: Bilirubin no greater than 2.0 mg/dL AST and ALT no greater than 4 times upper limit of normal (ULN) Albumin at least 3.0 g/dL PT and PTT no greater than 1.5 times ULN No liver failure Renal: Creatinine no greater than 1.7 mg/dL OR BUN no greater than 40 mg/dL No renal failure Other: Not pregnant or nursing Fertile patients must use effective contraception No serious infection No concurrent serious medical illness No allergy to penicillin or history of serious reaction to penicillamine No prior malignancy within the past 5 years except curatively treated carcinoma in situ or basal cell skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy for brain tumor No prior biologic therapy for brain tumor, including: Immunotoxins Immunoconjugates Antisense Peptide receptor antagonists Interferons Interleukins Tumor infiltrating lymphocytes Lymphokine activated killer cells Gene therapy No concurrent growth factors (e.g., filgrastim or epoetin alfa) Chemotherapy: No prior chemotherapy for brain tumor Endocrine therapy: Must be on stable corticosteroid regimen for at least 1 week (at least 5 days) No other prior hormonal therapy for brain tumor Radiotherapy: No prior radiotherapy for brain tumor Surgery: Recovered from prior surgery Other: No concurrent investigational agents No concurrent gold compounds (auronofin, gold sodium thiomalate) No concurrent herbal dietary supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1999-03; Primary Completion 2004-06 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Brem, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (9):
- United States (9):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Result] Brem S, Grossman SA, Carson KA, New P, Phuphanich S, Alavi JB, Mikkelsen T, Fisher JD; New Approaches to Brain Tumor Therapy CNS Consortium. Phase 2 trial of copper depletion and penicillamine as antiangiogenesis therapy of glioblastoma. Neuro Oncol. 2005 Jul;7(3):246-53. doi: 10.1215/S1152851704000869. PMID 16053699
- [Result] Brem S, Grossman SA, New P, et al.: Phase II study of penicillamine and reduction of copper, for angiosuppressive therapy of glioblastoma: preliminary safety and feasibility study. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A-666, 2000.